CLINICAL TRIAL: NCT05774262
Title: TELE-monitoring for Standard Pacemaker Implantation or Delayed Pacemaker Implantation After Autonomic/Electrophysiologic Evaluation and Cardioneuroablation for managEment of Functional atrioventriculaR Block - Randomized Controlled Study
Brief Title: Pacemaker Implantation Versus Cardioneuroablation for Functional Atrioventricular Block
Acronym: TELE-SPACER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American Heart of Poland (Other)
Responsible Party: Principal Investigator, Sebastian Stec, Clinical Professor, Principal Investigator, American Heart of Poland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/ABM/03/00035
Record Dates: First submitted 2023-02-17; First posted 2023-03-17 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Atrioventricular Block
Keywords: AVB; Pacemaker implantation; Cardioneuroablation; Cardiovascular autonomic testing (CAT); Telemedicine
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Intervention Model Description: multicenter, noncommercial, physician-initiated, proof-of-concept, prospective, randomized, controlled trial and registry
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - PACEMAKER (Active Comparator): Group A, n=50 patients aged 18-75 years with indications for elective PM implantation according to the 2021 ESC guidelines for cardiac pacing due to paroxysmal or persistent AVB with a positive results of atropine test.
  Group A is early elective pacemaker implantation (PM) strategy in functional AVB.
  Interventions: Procedure: Pacemaker implantation
- Group B - CARDIONEUROABLATION (Active Comparator): Group B, n=50 patients aged 18-75 years with indications for elective PM implantation according to the 2021 ESC guidelines for cardiac pacing due to paroxysmal or persistent AVB with a positive results of atropine test.
  Group B will undergo strategy of postponed/deferred PM implantation in functional AVB. Patients wil be implanted and monitored with ILR (in case of severe symptomatic AVB always the emergency system will be called). After cardiovascular autonomic testing (CAT), electrophysiological study (EPS), extra cardiac vagal nerve stimulation (ECVS) and cardioneuroablation will be performed. If CNA is succesful, pacemaker implantation will be cancelled. If CNA is unsuccessful, second session of CNA will be planned. In case of inefficient second attempt, patients will be referred for PM implantation. They will cross-over to PACEMAKER arm.
  Interventions: Procedure: Cardioneuroablation (CNA)

INTERVENTIONS:
Procedure: Pacemaker implantation — Elective pacemaker implantation (DDDR) for functional AVB according to the 2021 ESC Guidelines for Cardiac Pacing
  Arms: Group A - PACEMAKER
Procedure: Cardioneuroablation (CNA) — Experimental method; elective implantable loop recorder (ILR) and biatrial, binodal, atomically and electroanatomically guided CNA with extracardiac vagal nerve stimulation (ECVS) prior and after procedure monitoring (disappearance of ECVS-induced AVB with the goal of achieving post-procedure and maintaining a target heart rate > 50 beats per minute). CNA procedure is performed with radio-frequency generators and irrigated catheters and with support of 3D-electroanatomic mapping system.
  CNA group will receive external ECG recorders. The major reason for external ECG recorders is to provide documentation of clinical AVB, as well as monitoring of patients before and after CNA (or PM implantation, if accepted). In case of severe AVB symptoms always the emergency system will be called.
  Arms: Group B - CARDIONEUROABLATION

SUMMARY:
The TELE-SPACER study is a multicenter, noncommercial, physician-initiated, proof-of-concept, prospective, randomized, controlled, unblinded clinical trial and registry designed to compare two methods of treatment of patients with functional Atrio-Ventricular Block (AVB): the guidelines-recommended elective pacemaker (PM) therapy vs cardiovascular autonomic tests (CAT), electrophysiologic assessment (EPS) with referral to cardioneuroablation (CNA) and reevaluation of indications for PM therapy.

The main questions TELE-SPACER aims to answer are:

* Can the investigators successfully treat functional AVB without implantable device (PM)?
* Can the investigators prove the feasibility and safety and demonstrate non-inferiority of CNA procedure in patients with functional AVB, avoiding long-term permanent pacing, its limitations, complications and costs ?

The TELE-SPACER trial will validate the European Society of Cardiology (ESC) recommendations (level C of evidence: expert opinion) for elective PM implantation and will introduce CNA as effective treatment in the functional AVB patient population.

Functional AVB - defined as a persistent or paroxysmal AVB with a positive results of atropine test

DETAILED DESCRIPTION:
TELE-SPACER trial will enroll a minimum of 100 participants, males and females, 18-75 years old: 1) with indications for elective PM implantation due to atrioventricular block (AVB) according to 2021 ESC guidelines on cardiac pacing; 2) who had positive atropine tests. Participants will be randomized into two groups - either optimized guideline-recommended PM therapy (group A, n=50) or reevaluation for PM therapy after CAT/EPS and experimental procedure CNA (group B, n=50). Participants who will choose to opt-out of randomization will be included in the registry (group C) and will undergo patient-tailored intervention through shared decision-making with a possibility of either PM implantation, CNA or observation only. The registry is expected to include up to 200 participants.

Patient enrollment time is anticipated to last 2 years. Recruitment will take place in four study sites, in two distinct phases. First, the investigators will identify potential participants with AVB and a positive atropine test, confirming significant dependence of heart rhythm and conduction on the vagus nerve (hyperactivity of vagus nerve). Their medical records will be analyzed by the Scientific Committee (symptoms evaluation, physical examination, documentation of AVB). In the second phase eligible participants will be invited by the investigator to participate in the trial during medical consultation. After explanations describing the study protocol, including the risk and benefits, they will sign the written informed consent to participate in the study or will choose to opt-out of randomization to be included in the registry only (group C). Informed consent will be obtained only if it is clear that the patient truly understands the nature of the study. Alternatively, the patient will be encouraged to take a copy of the consent form home to contemplate enrolment in the study. Only participants who voluntarily consent will be included. Participants will be able to withdraw at any time without compromising their medical care.

Paricipants will be randomized in 1:1 allocation to either group A or group B. Randomization will be performed centrally and assigned automatically to each patient via internet. The randomization list will be blocked per center, with randomly varying block sizes of 2 and 4. The centers will not be aware of the block sizes. The PM implantation and treatment allocation will not be blinded to the patient or follow-up physician. Participants in either arm of the study will be followed-up at regular intervals for a minimum of 12 months. During the 12-month study duration, the use of effective contraception will be recommended for women of child-bearing age.

The period of the screening and randomization visit will last from 0 to 7 days, and the qualification for elective PM implantation (group A) or elective loop recorder monitoring/CAT/EPS (group B) and subsequent therapeutic decisions (CNA, DDDR, other treatment based on the test result) from 0 to 4 weeks. Parameter analysis baseline, including ECG telemonitoring, QOL and symptoms, will take place at randomization (0 months), 3, 6 and 12 months. Participants will be assessed using cardiovascular autonomic testing (CAT) with telemedical registration at 6 and 12 months. All measured parameters, as well as demographic and clinical data will be recorded in the study database.

Participants in group A (PM, n = 50) will receive care on the basis of the 2021 ESC Guidelines on Cardiac Pacing Recommendations. They will be implanted with PM (DDD pacemaker or its modification as HBP/LBBAP - His-Purkinje or left bundle branch area pacing) and will be monitored with external ECG recorder (certified medical devices of at least class IIa) with telemonitoring. Group B participants (CNA, n = 50) will be implanted with implantable loop recorder (ILR) device (Biotronik, Biomonitor 3m), also with remote tele-monitoring, with the same thresholds for automatic episode recording. As part of telemonitoring system, all participants will receive in the period before the procedure a dedicated telemonitoring kit consisting of a portable ECG device and a tablet with a sim card for network connection. This telemonitoring kit will enable regular self-testing, symptom reporting and interactive, objective telemedicine consultations. Participants will be provided with 24/7 contact with medical staff in the telemonitoring center specialized in cardiac arrhythmias and implantable device monitoring. The major reason for ECG recording is to provide ECG documentation of clinical AVB, as well as monitoring of participants before and after CNA (or PM implantation, if accepted). In case of severe AVB, the emergency system will always be called.

Participants in group B will be referred for EPS and ECVS (extracardiac vagal nerve stimulation) with the possibility of simultaneous CNA after exclusion of advanced and occult distal AVBs. Once the effectiveness of the CNA is confirmed, the patient will be further monitored. If CNA is not succesful and/or its immediate effectiveness is not confirmed (meeting the ESC criteria for pacemaker implantation after CNA), the patient will be referred for pacemaker implantation and will cross-over into group A.

CNA will be performed in group B under general anesthesia by experienced operators (at least 25 CNA procedures preformed). After EPS, a biatral, binodal, anatomically guided CNA will be performed under ECVS guidance, with a demonstration of the vagal reflex (complete asystole or AVB with atrial pacing) at the onset of the CNA and its complete disappearance after a successful CNA. Additional ablation substrates will also be allowed and performed.

Participants included in the registry (group C) will undergo an individually tailored intervention through shared decision making (SDM) with the option of implantation of PM (subgroup CA), CNA (subgroup CB) or observation only (subgroup C0).

All participants participating in the study and registry will be asked to complete questionnaires on health-related quality of life (EQ-5D-5L, SF-36), symptoms of bradycardia (VAS), fatigue (MFIS), depression (HADS-M) and sleep (ESS, AIS-8) at 0, 6, 12 months.

The safety of the interventions will be assessed on a monthly basis (telemedicine and standard follow-up visits), with monitoring of major adverse cardiovascular events (MACE). All events will be resolved by the Central Investigation Safety Committee, which does not include members of the Investigation Steering Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study
2. Age 18-75
3. Indication (at least one) of the European Society of Cardiology (ESC) for elective pacemaker implantation due to isolated (without sinus node dysfunction and bundle branch block) paroxysmal, persistent or reflex atrioventricular block:

   1. Symptomatic first degree AVB (above 300 msec). Class IIaC
   2. Symptomatic Mobitz type I second degree AVB. Class IIaC
   3. AVB 2:1, even asymptomatic, but not during sleep. Class IIaC
   4. Mobitz II type advanced 2nd degree AVB or complete block (3rd degree AVB). Class IC
   5. Advanced AVB during AF regardless of symptoms, but not during sleep. Class IC
   6. Reflex syncope in patients over 40 years of age with documented pauses within the AVB mechanism, symptomatic (>3 sec) or asymptomatic >6 sec. Class IC
   7. Reflex syncope in patients over 40 years of age with documented pauses within AVB mechanism in the course of sick sinus syndrome (CSS). Class IC
   8. Reflex syncope in patients over 40 years of age with documented pauses within AVB mechanism during tilt test. Class IC

Exclusion Criteria:

1. Implanted pacemaker/ICD/CRT
2. Sinus node dysfunction with indication for pacemaker implantation
3. Planned ablation of the atrioventricular junction
4. Severe prolonged bradycardia in advanced AVB requiring intravenous drugs and temporary pacing
5. Status post cardiac surgery
6. Acute myocardial infarction and heart failure (not related to bradycardia)
7. Status post percutaneous valvular intervention or ablation
8. Acute infection or any other accompanying disease which is contraindication to percutaneous procedures and/or implantation of a pacemaker
9. Pregnancy, nursing or planned pregnancy within 12 months
10. Decompensated chronic diseases (endocrine disorders, electrolyte disorders, etc.)
11. Advanced cardiomyopathies with indication for ICD implantation in primary or secondary prevention of sudden cardiac death (SCD)
12. Advanced ventricular arrhythmias with indication for ICD implantation in primary or secondary prevention of SCD
13. Persistent right or left bundle branch block
14. Musculoskeletal diseases with separate indications for pacemaker implantation
15. Contraindications to the procedures used in the study
16. The presence of a mental illness or limitation of cognitive functions that prevent independent participation in the study, including the use of telemedicine services
17. Any abnormality found that is considered by the Principal Investigator a contraindication to participate in the stidy due to data interpretation or safety issue

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of CNA in the treatment of AVB in comparison to PM therapy within 12 months of PM implantation/CNA procedure. | 12 months
  This is objective endpoint examining the onset of AVB episodes after PM/CNA. It will specify the number of pauses > 3.0 s in the ECG external recorder for group B (occurrence of > 1 pause or the need for earlier (0-12 months) PM implantation will be an indicator of the failure of the CNA procedure), assuming the presence of PM stimulation in group A at the level between 93-100% (equates to the continued duration of the AVB treated with PM).

SECONDARY OUTCOMES:
Occurrence of MACE (major advers cardiac events) | at 0, 3, 6, 12 months
  MACE are defined as peri-procedural and long-term complications: death, stroke, myocardial infarction, pericardial effusion requiring drainage, AVB, venous thrombosis, infection, hemorrhage, hematoma, fistula, pseudoaneurysm, surgical intervention
Assessment of the effect of CNA and PM implantation on AVB symptoms based on based on VAS (Visual Analog Scale) | 0, 3, 6, 12 months
  VAS (Visual Analog Scale) indicates the general health status with100 indicating the best health, 0 indicating the worst health status.
Assessment of the effect of CNA and PM implantation on health-related quality of life (QOL) based on questionaire EQ-5D-5L | 0, 6, 12 months
  EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is scored on a scale of 1-5 ponts, that describes the patient's health state. The maximum score of 1 indicates the best health state, higher scores indicate more severe or frequent problems.
Assessment of the effect of CNA and PM implantation on health-related quality of life (QOL) based on questionaire SF-36 | 0, 6, 12 months
  SF-36 questionnaire consists of 36 questions that are distributed across eight scales. Each scale is directly transformed into 0-100 scale. The lower the score the more disability, the higher the score the less disability.
Assessment of the effect of CNA and PM implantation on fatique based on Modified Fatigue Impact Scale (MFIS) | 0, 6, 12 moths
  MFIS is a validated, standardized, 21-item questionnaire, which provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. Total scores range from 0-84. The lower the score the less fatigue, the higher the score the more fatigue impairs physical, cognitive, and psychosocial functioning.
Assessment of the effect of CNA and PM implantation on depression/anxiety based on Modified Hospital Anxiety and Depression Scale (HADS-M) | 0, 6, 12 months
  HADS-M is a validated, standardized 16-item questionnaire to evaluate the association between anxiety and depression and the degree of illness acceptance in patients. Total scores range from 0-64. Higher scores indicate a greater degree of anxiety or depression.
Assessment of the effect of CNA and PM implantation on sleep disorders based on questionaire Epworth Sleep Scale (ESS) | 0, 6, 12 months
  The ESS score is a standardized, validated 8-item questionnaire (with scores 0-3 each). The total score can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life.
Assessment of the effect of CNA and PM implantation on sleep disorders based on Athens Insomnia Scale-8 (AIS-8) | 0, 6, 12 months
  AIS-8 is a standardized, validated questionnaire assessing 8 factors related to nocturnal sleep and daytime dysfunction, which are rated on a 0-3 scale. The sleep is evaluated from the cumulative score of all factors and reported as an individual's sleep outcome. Higher score indicates more sleep disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian M Stec, MD, PhD, Principal Investigator — American Heart of Poland; Edyta Stodolkiewicz-Nowarska, MD, PhD, Study Director — American Heart of Poland; Krzysztof Milewski, MD, PhD, Study Chair — American Heart of Poland
Locations (2):
- Poland (2):
  - American Heart of Poland, Dąbrowa Górnicza
  - American Heart of Poland, Mielec

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: Requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
  Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact PI smstec@wp.pl
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: De-identified individual participant level data and measurements including tables, figures, and appendices or supplementary material that support the results presented in a manuscript.
  Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact PI smstec@wp.pl

REFERENCES:
- [Background] Brignole M, Moya A, de Lange FJ, Deharo JC, Elliott PM, Fanciulli A, Fedorowski A, Furlan R, Kenny RA, Martin A, Probst V, Reed MJ, Rice CP, Sutton R, Ungar A, van Dijk JG; ESC Scientific Document Group. 2018 ESC Guidelines for the diagnosis and management of syncope. Eur Heart J. 2018 Jun 1;39(21):1883-1948. doi: 10.1093/eurheartj/ehy037. No abstract available. PMID 29562304
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Shen WK, Sheldon RS, Benditt DG, Cohen MI, Forman DE, Goldberger ZD, Grubb BP, Hamdan MH, Krahn AD, Link MS, Olshansky B, Raj SR, Sandhu RK, Sorajja D, Sun BC, Yancy CW. 2017 ACC/AHA/HRS Guideline for the Evaluation and Management of Patients With Syncope: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Circulation. 2017 Aug 1;136(5):e60-e122. doi: 10.1161/CIR.0000000000000499. Epub 2017 Mar 9. No abstract available. PMID 28280231
- [Background] Klank-Szafran M, Stec S, Sledz J, Janion M. [Radiofrequency ablation and cardioneuroablation for AVNRT and atrioventricular block]. Kardiol Pol. 2010 Jun;68(6):720-4. Polish. PMID 20806214
- [Background] Aksu T, Guler TE, Bozyel S, Ozcan KS, Yalin K, Mutluer FO. Cardioneuroablation in the treatment of neurally mediated reflex syncope: a review of the current literature. Turk Kardiyol Dern Ars. 2017 Dec;45(1):33-41. doi: 10.5543/tkda.2016.55250. PMID 28106018
- [Background] Baysal E, Guler TE, Gopinathannair R, Bozyel S, Yalin K, Aksu T. Catheter Ablation of Atrioventricular Block: From Diagnosis to Selection of Proper Treatment. JACC Case Rep. 2020 Sep 15;2(11):1793-1801. doi: 10.1016/j.jaccas.2020.07.050. eCollection 2020 Sep. PMID 34317058
- [Background] Aksu T, Gopinathannair R, Bozyel S, Yalin K, Gupta D. Cardioneuroablation for Treatment of Atrioventricular Block. Circ Arrhythm Electrophysiol. 2021 Sep;14(9):e010018. doi: 10.1161/CIRCEP.121.010018. Epub 2021 Sep 1. PMID 34465122
- [Background] Wileczek A, Polewczyk A, Kluk M, Kutarski A, Stec S. Ultrasound-guided imaging for vagus nerve stimulation to facilitate cardioneuroablation for the treatment of functional advanced atrioventricular block. Indian Pacing Electrophysiol J. 2021 Nov-Dec;21(6):403-406. doi: 10.1016/j.ipej.2021.06.008. Epub 2021 Jun 26. PMID 34186197
- [Background] Josiak K, Stec S, Zysko D, Skonieczny B, Kosior J, Sledz J, Wilczek A, Stodolkiewicz-Nowarska E, Biel B, Szymkiewicz P, Skoczynski P, Karbarz D, Ludwik B, Banasiak W, Jagielski D. Safety and efficacy of His bundle pacing validated by extracardiac vagal nerve stimulation (HIS-STORY). Cardiol J. 2022;29(4):698-701. doi: 10.5603/CJ.a2022.0053. Epub 2022 Jun 15. No abstract available. PMID 35703044
- [Background] Reichert A, Wileczek A, Stec S. Cardioneuroablation for the effective treatment of recurrent vasovagal syncope to restore driving abilities. Kardiol Pol. 2022;80(11):1158-1160. doi: 10.33963/KP.a2022.0189. Epub 2022 Aug 10. No abstract available. PMID 35946179
- [Background] Gajda R, Knechtle B, Gebska-Kuczerowska A, Gajda J, Stec S, Krych M, Kwasniewska M, Drygas W. Amateur Athlete with Sinus Arrest and Severe Bradycardia Diagnosed through a Heart Rate Monitor: A Six-Year Observation-The Necessity of Shared Decision-Making in Heart Rhythm Therapy Management. Int J Environ Res Public Health. 2022 Aug 19;19(16):10367. doi: 10.3390/ijerph191610367. PMID 36012002
- [Result] Pachon JC, Pachon EI, Pachon JC, Lobo TJ, Pachon MZ, Vargas RN, Jatene AD. "Cardioneuroablation"--new treatment for neurocardiogenic syncope, functional AV block and sinus dysfunction using catheter RF-ablation. Europace. 2005 Jan;7(1):1-13. doi: 10.1016/j.eupc.2004.10.003. PMID 15670960
- [Result] Pachon JC, Pachon EI, Cunha Pachon MZ, Lobo TJ, Pachon JC, Santillana TG. Catheter ablation of severe neurally meditated reflex (neurocardiogenic or vasovagal) syncope: cardioneuroablation long-term results. Europace. 2011 Sep;13(9):1231-42. doi: 10.1093/europace/eur163. Epub 2011 Jun 28. PMID 21712276
- [Result] Pachon M JC, Pachon M EI, Santillana P TG, Lobo TJ, Pachon CTC, Pachon M JC, Albornoz V RN, Zerpa A JC. Simplified Method for Vagal Effect Evaluation in Cardiac Ablation and Electrophysiological Procedures. JACC Clin Electrophysiol. 2015 Oct;1(5):451-460. doi: 10.1016/j.jacep.2015.06.008. Epub 2015 Aug 21. PMID 29759475
- [Result] Yao Y, Shi R, Wong T, Zheng L, Chen W, Yang L, Huang W, Bao J, Zhang S. Endocardial autonomic denervation of the left atrium to treat vasovagal syncope: an early experience in humans. Circ Arrhythm Electrophysiol. 2012 Apr;5(2):279-86. doi: 10.1161/CIRCEP.111.966465. Epub 2012 Jan 24. PMID 22275485
- [Result] Hu F, Zheng L, Liang E, Ding L, Wu L, Chen G, Fan X, Yao Y. Right anterior ganglionated plexus: The primary target of cardioneuroablation? Heart Rhythm. 2019 Oct;16(10):1545-1551. doi: 10.1016/j.hrthm.2019.07.018. Epub 2019 Jul 19. PMID 31330187
- [Result] Sun W, Zheng L, Qiao Y, Shi R, Hou B, Wu L, Guo J, Zhang S, Yao Y. Catheter Ablation as a Treatment for Vasovagal Syncope: Long-Term Outcome of Endocardial Autonomic Modification of the Left Atrium. J Am Heart Assoc. 2016 Jul 8;5(7):e003471. doi: 10.1161/JAHA.116.003471. PMID 27402231
- [Result] Aksu T, Golcuk E, Yalin K, Guler TE, Erden I. Simplified Cardioneuroablation in the Treatment of Reflex Syncope, Functional AV Block, and Sinus Node Dysfunction. Pacing Clin Electrophysiol. 2016 Jan;39(1):42-53. doi: 10.1111/pace.12756. Epub 2015 Oct 26. PMID 26411271
- [Result] Osorio TG, Paparella G, Stec S, Chierchia GB, de Asmundis C. Cardiac parasympathetic modulation in the setting of radiofrequency ablation for atrial fibrillation. Arch Med Sci. 2019 Apr 26;17(6):1716-1721. doi: 10.5114/aoms.2019.84717. eCollection 2021. PMID 34900053
- [Result] Piotrowski R, Baran J, Kulakowski P. Cardioneuroablation using an anatomical approach: a new and promising method for the treatment of cardioinhibitory neurocardiogenic syncope. Kardiol Pol. 2018;76(12):1736-1738. doi: 10.5603/KP.a2018.0200. Epub 2018 Oct 19. No abstract available. PMID 30338504
- [Result] Pachon-M EI, Pachon-Mateos JC, Higuti C, Santillana-P TG, Lobo T, Pachon C, Pachon-Mateos J, Zerpa J, Ortencio F, Amarante RC, Silva RF, Osorio TG. Relation of Fractionated Atrial Potentials With the Vagal Innervation Evaluated by Extracardiac Vagal Stimulation During Cardioneuroablation. Circ Arrhythm Electrophysiol. 2020 Apr;13(4):e007900. doi: 10.1161/CIRCEP.119.007900. Epub 2020 Mar 19. PMID 32188285